CLINICAL TRIAL: NCT03272802
Title: Treatment Effect of Edaravone in Patients With Amyotrophic Lateral Sclerosis (ALS) in a Representative Iranian Population
Brief Title: Treatment Effect of Edaravone in Patients With Amyotrophic Lateral Sclerosis (ALS)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Alireza Eishi Oskouei, MD, Isfahan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Isfahan ALS Registery
Record Dates: First submitted 2017-09-02; First posted 2017-09-06 (Actual); Last update posted 2019-03-27 (Actual); Status verified 2019-03

CONDITIONS: Neuromuscular Diseases
Keywords: Amyotrophic Lateral Sclerosis; Edaravone
MeSH Terms: conditions — Neuromuscular Diseases; Amyotrophic Lateral Sclerosis | interventions — Edaravone; Riluzole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): ALS patients who receive the usual treatment option (Riluzole) for this disease and Edaravone. Instructions:
  1. Tab. Rilutek 50 mg PO q12hr on empty stomach.
  2. Amp. Edaravone 60 mg per day IV infusion (in normal saline during 1 hour) for 14 days in the first 28 day cycle.
  3. Amp. Edaravone 60 mg per day IV infusion (in normal saline during 1 hour) for 10 days in the following 28 day cycles after the first cycle (for 11 cycles).
  Interventions: Drug: Edaravone; Drug: Riluzole
- Control group (Active Comparator): ALS patients who receive the usual treatment option (Riluzole) for this disease.
  Instructions:
  1. Tab. Rilutek 50 mg PO q12hr on empty stomach.
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Edaravone — Edaravone is a free radical scavenger. this drug showed desirable effects like slowing decline of physical function by 33 percent in previous studies.
  Other Names: Radicut; RADICAVA
  Arms: Case group
Drug: Riluzole — Riluzole is a treatment option for amyotrophic lateral sclerosis. The occurrence of ventilator-dependence or tracheostomy is delayed in selected patients who treated with this drug.
  Other Names: Rilutek; Teglutik

SUMMARY:
Amyotrophic Lateral Sclerosis (ALS) is a neurodegenerative disease that causes the death of 30,000 affected individual every year. Complex nature and unknown pathogenesis of this disease are 2 major reasons for failure of therapeutic interventions. Edaravone is a free radical scavenger that slows down functional decline and prevents from disease progression in ALS patients. FDA newly approved this drug in these patients (2017/5/5). In this study, investigators aimed to assess the treatment effect of this newly approved drug in patients with ALS in a representative Iranian population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as definite or probable ALS according to El Escorial Criteria.
2. ALS patients who are graded as mild or moderate according to ALS Health State Scale.
3. Forced vital capacity of at least 80%
4. Desire of the patient to participate in this study and Signing Written Informed Consent.

Exclusion Criteria:

1. Incidence of drug's side effects that requires discontinuation of the drug (Edaravone's side effects: Acute kidney injury, Acute allergic reactions, DIC, Thrombocytopenia, Leukopenia).
2. Desire of the patient to discontinue participating in this study.
3. the patient starts another drug or herb for ALS during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-03-16 (Actual); Primary Completion 2019-03-16 (Estimated); Study Completion 2019-09-16 (Estimated)

PRIMARY OUTCOMES:
Functional evaluation of patient's muscle strength. | At the time of enrolling the patient to study, and then every 3 moths in the following period of 1 year.
  Manual Muscle Testing (MMT) will be used to evaluate functional muscle strength. This procedure evaluates the strength of some proximal and distal muscles of each limb and also the neck region.
functional status of the patient. | At the time of enrolling the patient to study, and then every 3 moths in the following period of 1 year.
  Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) will be used to evaluate functional status of the patient.
Quality of life in the patients | At the time of enrolling the patient to study, and then every 3 moths in the following period of 1 year.
  Amyotrophic Lateral Sclerosis Assessment Questionnaire (ALSAQ-40) will be used to assess Quality of life in the patients. The Persian version of this questionare will be used in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- EMG Department, Alzahra Hospital, Isfahan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shamshiri H, Fatehi F, Davoudi F, Mir E, Pourmirza B, Abolfazli R, Etemadifar M, Harirchian MH, Gharagozli K, Ayromlou H, Basiri K, Zamani B, Rohani M, Sedighi B, Roudbari A, Delavar Kasmaei H, Nikkhah K, Ranjbar Naeini A, Nafissi S. Amyotrophic lateral sclerosis progression: Iran-ALS clinical registry, a multicentre study. Amyotroph Lateral Scler Frontotemporal Degener. 2015;16(7-8):506-11. doi: 10.3109/21678421.2015.1074698. Epub 2015 Oct 5. PMID 26437387
- [Background] Abe K, Itoyama Y, Sobue G, Tsuji S, Aoki M, Doyu M, Hamada C, Kondo K, Yoneoka T, Akimoto M, Yoshino H; Edaravone ALS Study Group. Confirmatory double-blind, parallel-group, placebo-controlled study of efficacy and safety of edaravone (MCI-186) in amyotrophic lateral sclerosis patients. Amyotroph Lateral Scler Frontotemporal Degener. 2014 Dec;15(7-8):610-7. doi: 10.3109/21678421.2014.959024. Epub 2014 Oct 6. PMID 25286015
- [Background] Writing Group; Edaravone (MCI-186) ALS 19 Study Group. Safety and efficacy of edaravone in well defined patients with amyotrophic lateral sclerosis: a randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2017 Jul;16(7):505-512. doi: 10.1016/S1474-4422(17)30115-1. Epub 2017 May 15. PMID 28522181
- [Derived] Eishi-Oskouei A, Basiri K. Safety and efficacy of edaravone in well-defined Iranian patients with amyotrophic lateral sclerosis: A parallel-group single-blind trial. Curr J Neurol. 2021 Jan 4;20(1):1-7. doi: 10.18502/cjn.v20i1.6373. PMID 38011420